[Type the document title]
Effectiveness of Early Oral
Feeding vs Traditional NPO
Protocol in Reduction of
Postoperative Complications
In Emergency Abdominal
Surgeries

[Type the document subtitle]

8/10/2018 Dr.Ayesha Masood Windows User



# REGISTRATION & RESEARCH CELL

### RESEARCH EVALUATION UNIT

Ref No: CPSP/REU/SGR-2016-126-8181 Dated: August 10, 2018

For quick and effective communication please send us your email address

Dr. AYESHA MASOOD HOUSE NO.F 214/5, STREET NO.8, PHASE-II, OFFICERS COLONY, WAH CANTT Phone No: 0514532119, -

Dear Doctor,

Please refer to your synopsis of Dissertation / Article titled:

"EFFECTIVENESS OF EARLY ORAL FEEDING VS TRADITIONAL NPO PROTOCOL IN REDUCTION OF POST OPERATIVE COMPLICATIONS IN EMERGENCY ABDOMINAL SURGERIES."

This is to inform you that your synopsis of Dissertation/Article has been <u>APPROVED</u>. Please note that the changes advised in the attached documents are to be incorporated in the dissertation.

#### Please note:

- The Research study should be commenced after the approval of synopsis, with the attached conditions fulfilled in the dissertation.
- The dissertation must be submitted at least six months prior to Examination (dates on website).

The following documents must be submitted with the dissertation at the time of submission.

- 1. Application form for submission of dissertation & data.
- 2. Experience Proforma (Certificate).
- 3. Dissertation data sheets.
- Copy of the approved synopsis.
- 5. Supervisor's signed and stamped covering letter.

Please quote above Reference No. in all future correspondence.

Yours sincerely,

2

DR. MUHAMMAD TARIQ KARIM

Senior Lecturer,

Research Evaluation Unit, CPSP

College of Physicians and Surgeons Pakistan

**BACKGROUND**: Enhanced recovery after surgery (ERAS) protocols have been widely studied in elective abdominal surgeries and have shown better outcomes. However the utility of these protocols in emergency abdominal surgeries has not been widely investigated.

**OBJECTIVE**: To study the outcomes of application of ERAS protocols in patients undergoing perforated duodenal ulcers repairs in emergency abdominal surgeries.

**DESIGN:** Randomized Controlled Trial.

**PLACE AND DURATION OF STUDY:** This randomized controlled trial was conducted in Surgical Unit 1 BBH from August 2018 to December 2019.

**METHODS**: Patients presenting to the emergency department with peritonitis secondary to suspected perforated duodenal ulcer were admitted. Total sample size of the study was 36 patients. Patients were randomly divided in two groups. Group A consisted of early oral feeding group and group B consisted of traditional postoperative care group. Outcome results studied were the length of hospital stay, duodenal repair site leak, severity of pain (VAS score) and duration of postoperative ileus. Results were analysed on SPSS version 20 and chisquare and independent t-test were applied

# **Statistical Analysis Plan:**

All data was entered and analyzed using SPSS (statistical package for social sciences) version 20. The categorical values like gender and types of surgery were expressed as frequency or percentages. The quantitative variables like age, post operative pain and length of hospital stay, days of return of bowel function were expressed as mean or standard deviation. Student t test was applied to compare hospital stay, days of return of bowel function and pain score between two groups. Effect modifiers like age and gender along with type of surgery were controlled by stratification and post stratification student t test was applied. P value of<0.05 would be considered statistically significant

# PATIENT CONSENT FORM

Department Of Surgery Unit-1 Benazir Bhutto Hospital, Rawalpindi

## EFFECTIVENESS OF EARLY ORAL FEEDING VS TRADITIONAL NPO PROTOCOL IN REDUCTION OF POST OPERATIVE COMPLICATIONS IN EMERGENCY ABDOMINAL **SURGERIES**

| oroject. I am giving consent to ordinate and disadvantages of over Dr | is fully informed about the research enroll myself in this research as a subject. The the interventions are clearly explained to me of any mishap or adverse effect of intervention, tal staff will be responsible and I will not sue |
|---|---|
| Name and signature of Patient Diagnosis | |
| Name and signature of Doctor | |
| Date | |